CLINICAL TRIAL: NCT04986488
Title: Incidence And Predictors of Delirium After Cardiac Surgery; A Prospective Observational Cohort Study From a Single Tertiary Referral Centre
Brief Title: INCIDENCE OF Delirium After Cardiac SURGERY Surgery
Status: Completed | Type: Observational
Sponsor: Shahid Gangalal National Heart Centre (Other)
Responsible Party: Principal Investigator, Smriti Mahaju Bajracharya,MD, Registrar in cardiac anesthesiology and critical care, Shahid Gangalal National Heart Centre
Other Study IDs: SGNHC 2
Record Dates: First submitted 2021-07-12; First posted 2021-08-02 (Actual); Last update posted 2021-08-02 (Actual); Status verified 2021-07

CONDITIONS: Delirium
Keywords: delirium;post-cardiac surgery;adults
MeSH Terms: conditions — Delirium

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Without delirium
- With delirium

SUMMARY:
Delirium is a common problem that occurs after cardiac surgery. The incidence of delirium after cardiac surgery is estimated to be 26-52%, with a significant percentage being hypoactive delirium1-4.Postoperative delirium has been associated with higher hospital costs, longer lengths of hospital stay, increased likelihood of institutionalization, increased risk for dementia, and increased morbidity and mortality.5-7 .

The overall purpose of this study was to determine the incidence and perioperative factors that predispose to cause delirium in postoperative cardiac surgery patients in our ICU

ELIGIBILITY:
Inclusion Criteria:

* Patients 18 years old and older of both sexes
* Patients who signed an informed consent
* Patients scheduled for cardiac surgery with extracorporeal circulation (coronary-artery bypass grafting (CABG), cardiac valve replacement (CVR), combined CABG + CVR, excision of cardiac myxoma)

Exclusion Criteria:

* Patients who refused to participate before or after operation;
* Patients in poor general condition;
* Patients with preoperative dementia, delirium or illiterate, psychiatric or mental disorder (epilepsy, schizophrenia, depression);
* Patients who died intraoperatively or within the first 6 hours after the procedure.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients 18 years old and older of both sexes who are undergoing cardiac surgery in a single centre
Sampling Method: Non-Probability Sample
Enrollment: 234 (Actual)
Dates: Start 2018-07-01 (Actual); Primary Completion 2018-12-30 (Actual); Study Completion 2018-12-30 (Actual)

PRIMARY OUTCOMES:
incidence and perioperative factors that predispose to cause delirium in postoperative cardiac surgery patients in our ICU | 6 months
  Incidence and perioperative risk factors that may predispose to delirium after cardiac surgery in our settings

SECONDARY OUTCOMES:
ICU stay and mechanical ventilation time | 6 months
  whetherICU stay in days and mechanical ventilation time in number of hours is affected by delirium

CONTACTS AND LOCATIONS:
Locations (1):
- Shahid Gangalal National Heart Center, Kathmandu, Nepal